CLINICAL TRIAL: NCT06416020
Title: Integrating MOUD in Nonmedical Community Settings (Better Together)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Howard University (Other)
Collaborators: University of Illinois at Chicago (Other); University of Miami (Other); National Institute on Drug Abuse (NIDA) (NIH); The Emmes Company, LLC (Industry); University of Maryland (Other)
Responsible Party: Principal Investigator, Richard Schottenfeld, Professor and Chair, Department of Psychiatry, Howard University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIDA CTN Protocol 0144; UG1DA013720 (NIH)
Record Dates: First submitted 2024-04-19; First posted 2024-05-16 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Opioid Use Disorder
Keywords: MOUD; OUD; Buprenorphine
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine

STUDY DESIGN:
Intervention Model Description: A multisite hybrid Type 1 effectiveness-implementation randomized clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hub Clinic MOUD with buprenorphine only (HC-MOUD Only) (Active Comparator): Participants will receive MOUD with buprenorphine prescribed by providers based at participating hub clinics. MOUD treatment with buprenorphine will follow standard guidelines for induction and maintenance using a sublingual buprenorphine formulation. Hub clinic buprenorphine providers and participants may shift to long acting injection buprenorphine formulations after initial induction with sublingual buprenorphine. If telemedicine prescribing of MOUD with buprenorphine is part of the usual standard of care at the clinic, participants assigned to HC-MOUD Only may be prescribed buprenorphine via telemedicine, following the clinic's usual guidelines. Participants may not receive telemedicine services at the community spokes or Recovery Guiding, which are available only to participants assigned to BTMOUD. All study participants, however, may have access to any services that are routinely provided as part of the MOUD with buprenorphine treatment-as-usual care in the hub clinic.
  Interventions: Behavioral: HC-MOUD Only
- Recovery Guiding / Better Together Medications for Opioid Use Disorder (BT-MOUD) procedures (Experimental): Better Together Medications for Opioid Use Disorder (BT-MOUD) includes HC-MOUD plus access to telemedicine provision of MOUD with buprenorphine at a nonmedical community organization spoke, plus manual-guided Recovery Guiding provided onsite at the spoke, and plus any other services available at the community organization spoke. Recovery Guiding is a manualized, highly structured, stepwise intervention that uses educational and behavioral tools to provide pragmatic guidance for patients beginning buprenorphine treatment and to address the key recovery misconceptions and dysfunctional behaviors that frequently interfere with recovery efforts of patients initiating medication for opioid use disorder (MOUD) treatment.
  Interventions: Behavioral: BT-MOUD with Buprenorphine

INTERVENTIONS:
Behavioral: HC-MOUD Only — MOUD with buprenorphine provided in a hub buprenorphine clinic
  Other Names: Hub Clinic MOUD with Buprenorphine
  Arms: Hub Clinic MOUD with buprenorphine only (HC-MOUD Only)
Behavioral: BT-MOUD with Buprenorphine — MOUD with buprenorphine provided by a hub buprenorphine provider either in the hub clinic or via telemedicine at a community hub; Recovery Guiding provided to participants
  Other Names: Better Together MOUD with Buprenorphine
  Arms: Recovery Guiding / Better Together Medications for Opioid Use Disorder (BT-MOUD) procedures

SUMMARY:
A multisite effectiveness-implementation study will be conducted in four sites to evaluate interventions to improve engagement and retention in MOUD with buprenorphine treatment persons with Opioid Use Disorder (OUD) in urban neighborhoods with high overdose rates. The investigators hypothesize that treatment with the Better Together Integrated Collaborative Community MOUD care model (BT-MOUD) will result in better retention in treatment than standard-of-care MOUD with buprenorphine provided in the hub buprenorphine clinic only (HC-MOUD Only) through 24 weeks following randomization. BT-MOUD provides MOUD with buprenorphine in nonmedical community-based settings via telemedicine from a hub buprenorphine clinic combined with Recovery Guiding, a manual guided coaching developed for this approach, provided onsite in the community organization.

DETAILED DESCRIPTION:
This multi-site hybrid Type 1 effectiveness-implementation study conducted in Washington, District of Columbia (DC), Chicago, Miami-Dade County and Baltimore will evaluate: 1) the effectiveness of providing MOUD with buprenorphine onsite (via telemedicine from a hub buprenorphine clinic) combined with Recovery Guiding in nonmedical community-based settings (the Better Together Integrated Collaborative Community MOUD care model - BT-MOUD) compared to standard-of-care MOUD with buprenorphine provided in the hub buprenorphine clinic only (HC-MOUD Only) and 2) BT-MOUD implementation barriers and facilitators. In the BT-MOUD intervention, community sites serve as "spokes" for telemedicine provision of MOUD by buprenorphine providers based in a "hub" buprenorphine clinic. A trained and supervised Recovery Guide with roots or connections with the community provides manual-guided Recovery Guiding on-site in the community site. Recovery Guiding includes psychoeducation (about OUD and effective buprenorphine MOUD) and behavioral counseling to promote engagement in MOUD with buprenorphine, retention in care, medication adherence, and behavioral change supportive of recovery. In HC-MOUD Only, participants will receive MOUD with buprenorphine and other available services in the hub buprenorphine clinic only. A Peer Outreach Specialist (POS) will assist with outreach and recruitment of all participants across conditions and with maintaining high rates of follow-up in research assessments. This study will test the hypothesis that BT-MOUD is more effective than HC-MOUD Only in retaining persons with OUD in MOUD with buprenorphine through six months post-randomization.

ELIGIBILITY:
Inclusion Criteria

1. Be 16 years of age or older
2. Has been newly prescribed MOUD with buprenorphine by a hub clinic provider no more than 10 days before the day of randomization or on the day of randomization [Note that the "start" of a "current, new treatment episode" of MOUD with buprenorphine is defined as the date MOUD with buprenorphine was prescribed by a hub clinic provider.]
3. Is willing and able to provide written informed consent
4. Is willing and able to provide reliable locator information to facilitate contacting the participant for research follow-up assessments
5. Speaks English well enough to be able to comprehend the study procedures and complete the assessments

Exclusion Criteria:

1. In the 30 days prior to receiving the prescription for MOUD with buprenorphine from the hub clinic provider, has either taken prescribed MOUD as an outpatient for more than 10 consecutive days OR received injectable MOUD that covers more than 10 consecutive days [Note that receipt of MOUD in a hospital, residential treatment, or carceral setting would not trigger exclusion.]
2. Plans to move out of the area or anticipate not being able to remain in the study for 6 months
3. Is currently in jail, prison, or other overnight facility as required by a court of law or have pending legal action that could prevent participation in study activities
4. Has been previously enrolled in CTN-0144 or CTN-0088 or is currently enrolled in another clinical trial for treatment of OUD

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2026-01-26 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Buprenorphine MOUD Treatment Retention | 0-168 days
  Duration of continuous participation in the hub clinic provided buprenorphine treatment

SECONDARY OUTCOMES:
Self-reported adherence to MOUD with buprenorphine | 0-168 days
  Number of days self-reported adherence to MOUD with buprenorphine assessed using timeline follow back (TLFB) Adherence to buprenorphine during the 168-day study period
Self-reported nonmedical opioid use | 0-168 days
  Number of days self-reported days of nonmedical opioid use, stimulant use, benzodiazepine use during the 168 study period
Self-reported nonmedical other drug use | 0-168 days
  Number of days self-reported other drug use
Urine Toxicology | Months 1,2 3,4,5,6
  Number of opioid-negative urine toxicology tests, ranging from 0 to 6.
Health-related quality of life (HRQOL) | Months 1,2 3,4,5,6
  Assess quality of life using the Health-related Quality of Life Health Related Quality of Life -4: Scores range from 1-5 for Q1, assessing overall health-related quality of life, and from 0-30 for Q2, Q3, and Q4 assessing physical health (Q2), mental health (Q3), and interference from health or mental health problems (Q4); higher scores indicate worse outcomes.
Patient Health Questionnaire Depression Scale | Months 1,2,3,4,5,6
  Assess depressive symptoms using Patient Health Questionnaire Depression Scale-8 (PHQ-8). Scores range from 0 to 24. Higher scores are indicators of greater depression severity.
Pharmacy Dispensed Buprenorphine | Months 1, 2, 3, 4, 5, 6
  Data regarding HUB clinic prescribed buprenorphine that is dispensed to the participant by a pharmacy will be obtained as part of the abstraction of data from electronic medical and pharmacy records.

CONTACTS AND LOCATIONS:
Overall Officials: Richard S Schottenfeld, MD, Principal Investigator — Howard University; Viviana Horigian, MD, MHA, Principal Investigator — University of Miami; Niranjan Karnik, MD, PhD, Principal Investigator — University of Illinois Chicago; Denise M. Scott, PhD, Study Director — Howard University
Locations (4):
- United States (4):
  - Howard University, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - University of Illinois- Chicago, Chicago, Illinois
  - University of Maryland, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: Yes
This study will comply with the NIH Policy for Data Management and Sharing (Notice Number: NOT-OD-21-013) (https://grants.nih.gov/grants/policy/data_sharing/data_sharing_guidance.htm) and for Helping to End Addiction Long-Term (HEAL) funded studies) the HEAL Public Access and Data Sharing Policy (https://www.nih.gov/research-training/medical-research-initiatives/heal initiative/research/heal public-access-data-sharing-policy)]. For more details on data sharing please visit https://datashare.nida.nih.gov/.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Datasets for Clinical Trials Network Protocol -144 (CTN-0144) will be available when either (1) the primary outcome paper has been accepted for publication, (2) the data has been locked for more than 18 months, or (3) the grant concludes; whichever comes first. The datasets will remain accessible via NIDA Data Share contingent on NIDA's continued support of the archive. To date, NIDA Data Share has not deleted any deposited data.
Access Criteria: Access to the scientific data generated from CTN-0144 will be controlled via a registration agreement for data use on the NIDA Data Share Website.
URL: https://datashare.nida.nih.gov/